CLINICAL TRIAL: NCT03067129
Title: An Open-Label, Multicenter Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Glecaprevir/Pibrentasvir in Pediatric Subjects With Genotypes 1-6 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Glecaprevir/Pibrentasvir in Pediatric Subjects With Genotypes 1-6 Chronic Hepatitis C Virus (HCV) Infection
Acronym: DORA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-123; 2016-004102-34 (EudraCT Number)
Expanded Access: NCT03123965 (Approved for marketing)
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C Virus; Glecaprevir; Pibrentasvir; Pharmacokinetic; Treatment naïve; Treatment experienced; Interferon (IFN); Pegylated interferon (pegIFN); Ribavirin (RBV); Sofosbuvir; Non-cirrhotic cirrhosis; Compensated (Child-Pugh A) cirrhosis
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Fibrosis | interventions — glecaprevir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Adult Formulation; 12 to < 18 years (Experimental): Adolescents aged 12 to < 18 years old received the adult formulation of glecaprevir (GLE)/pibrentasvir (PIB) 100 mg/ 40 mg co-formulated film-coated tablets for a once daily (QD) total dose of 300 mg/120 mg by mouth for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience.
  Interventions: Drug: Glecaprevir/Pibrentasvir Adult Formulation
- Cohort 2: Pediatric Formulation; 9 to < 12 years (Experimental): Children aged 9 to < 12 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience.
  The initial proposed dose for children 9 to < 12 years old (30 to < 45 kg) was GLE 200 mg + PIB 75 mg. After PK analysis from the first 6 enrolled participants the dose was adjusted to GLE 250 mg + PIB 100 mg.
  Interventions: Drug: Glecaprevir + Pibrentasvir Pediatric Formulation
- Cohort 3: Pediatric Formulation; 6 to < 9 years (Experimental): Children aged 6 to < 9 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience.
  The initial proposed dose for children 6 to < 9 years old (20 to < 30 kg) was GLE 160 mg + PIB 60 mg. After PK analysis from the first 6 enrolled participants the dose was adjusted to GLE 200 mg + PIB 80 mg.
  Interventions: Drug: Glecaprevir + Pibrentasvir Pediatric Formulation
- Cohort 4: Pediatric Formulation; 3 to < 6 years (Experimental): Children aged 3 to < 6 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience.
  The initial proposed dose for children 3 to < 6 years old (12 to < 20 kg) was GLE 120 mg + PIB 45 mg. After PK analysis from the first 5 enrolled participants the dose was adjusted to GLE 150 mg + PIB 60 mg.
  Interventions: Drug: Glecaprevir + Pibrentasvir Pediatric Formulation

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir Adult Formulation — Co-formulated film-coated tablet (100 mg/40 mg)
  Other Names: ABT-493/ABT-530; MAVYRET®
  Arms: Cohort 1: Adult Formulation; 12 to < 18 years
Drug: Glecaprevir + Pibrentasvir Pediatric Formulation — Film-coated pellets/granules (15.67%/8.25%) administered by mixing with a small amount (1-2 teaspoons) of a soft food vehicle, such as hazelnut spread, Greek yogurt, or peanut butter.
  Other Names: ABT-493/ABT-530
  Arms: Cohort 2: Pediatric Formulation; 9 to < 12 years; Cohort 3: Pediatric Formulation; 6 to < 9 years; Cohort 4: Pediatric Formulation; 3 to < 6 years

SUMMARY:
The objectives of this study are to assess the pharmacokinetics, safety, and efficacy of glecaprevir/pibrentasvir adult formulation in adolescents ages 12 to 17 years and a pediatric formulation of glecaprevir and pibrentasvir in children ages 3 to < 12 years.

DETAILED DESCRIPTION:
This was a multicenter study to evaluate the pharmacokinetics (PK), efficacy, and safety of glecaprevir (GLE) and pibrentasvir (PIB) treatment for 8, 12, or 16 weeks in hepatitis C virus (HCV) genotype 1 - 6 (GT1 - GT6)-infected pediatric participants 3 to < 18 years of age, with or without compensated cirrhosis, with or without human immunodeficiency virus (HIV) coinfection, who are either treatment-naïve (TN), treatment-experienced (TE) with pegylated interferon (pegIFN) with or without ribavirin (RBV), or TE with sofosbuvir (SOF) + RBV with or without pegIFN.

The study was divided into 2 parts, according to the formulation of GLE/PIB administered. Part 1 of the study enrolled HCV GT1 - GT6 infected adolescent participants into the 12 to < 18 years old age group who were willing to swallow the adult formulation of GLE/PIB (Cohort 1). Part 2 of the study enrolled HCV GT1 - GT6 infected pediatric participants divided into the 9 to < 12 (Cohort 2), 6 to < 9 (Cohort 3), and 3 to < 6 (Cohort 4) years old age groups, to receive the pediatric formulation of GLE + PIB. Part 1 enrolled first and once the pediatric formulation was available enrollment into Part 2 commenced, with each cohort enrolled in parallel.

In each cohort, the first group of participants were enrolled into an intense pharmacokinetics (IPK) portion to characterize the PK and safety in each age group, followed by enrollment into a non-IPK safety/efficacy portion. Study participants enrolled in the IPK portion must have been HIV-negative, treatment-naive, and have an identified HCV genotype. In the IPK portion the first approximately six participants received an initial proposed dose of GLE and PIB based on the child's weight and age at screening. PK samples from these participants were evaluated to determine if therapeutic efficacious exposures were attained, comparable to those of adults, and if any dose adjustments were needed. After the intensive PK analysis results for the first six participants were available, enrollment of the remaining IPK portion resumed with subsequent participants receiving an adjusted final dose as applicable. Additional participants may have been required for further intensive PK analysis per age cohort if therapeutic exposure targets were not achieved.

Enrollment into the non-IPK safety and efficacy portions began when the dosing recommendations per age group based on the PK and clinical data from the IPK analysis were ascertained.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus (HCV) infection demonstrated by positive anti-HCV antibody (Ab) and HCV ribonucleic acid (RNA) greater than or equal to 1000 International Unit (IU)/mL
* Subjects participating in the intense pharmacokinetic (IPK) part must have been HCV treatment-naive, with or without compensated cirrhosis (Child-Pugh A), human immunodeficiency virus type 1 (HIV-1) negative and must have had a Screening laboratory result indicating HCV genotype (GT) 1, 2, 3, 4, 5, or 6-infection.

Exclusion Criteria:

* Females who were pregnant or breastfeeding
* Positive test result for hepatitis B surface antigen (HbsAg) or positive test result for hepatitis B virus deoxyribonucleic acid (DNA)
* Participants with other known liver diseases
* Decompensated cirrhosis defined as: presence of ascites, history of variceal bleeding, lab values consistent with Child-Pugh class B or C cirrhosis

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (38):
- United States (15):
  - Univ of California San Francis /ID# 158002, San Francisco, California
  - Childrens Hospital Colorado /ID# 157996, Aurora, Colorado
  - CT Childrens Medical Ctr, US /ID# 158639, Hartford, Connecticut
  - UF Hepatology Research at CTRB /ID# 158008, Gainesville, Florida
  - Advent Health /ID# 166022, Orlando, Florida
  - Indiana University /ID# 158001, Indianapolis, Indiana
  - Boston Childrens Hospital /ID# 157988, Boston, Massachusetts
  - Boston Medical Center /ID# 157997, Boston, Massachusetts
  - Columbia Univ Medical Center /ID# 158000, New York, New York
  - UNC Health Care /ID# 157991, Chapel Hill, North Carolina
  - Cincinnati Childrens Hosp Med /ID# 158007, Cincinnati, Ohio
  - Children's Hospital of Philadelphia /ID# 158003, Philadelphia, Pennsylvania
  - Child Hosp of Pittsburgh,PA /ID# 158004, Pittsburgh, Pennsylvania
  - Monroe-Carell Jr. Children's H /ID# 169037, Nashville, Tennessee
  - Baylor College of Medicine /ID# 157989, Houston, Texas
- Belgium (2):
  - Cliniques Universitaires Saint Luc /ID# 162173, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Leuven /ID# 162174, Leuven
- Canada (3):
  - Alberta Children's Hospital /ID# 163449, Calgary, Alberta
  - Stollery Children's Hospital /ID# 163450, Edmonton, Alberta
  - Hospital for Sick Children /ID# 163448, Toronto, Ontario
- Germany (3):
  - Universitatsklinikum Freiburg /ID# 165187, Freiburg im Breisgau, Baden-Wurttemberg
  - Charite Universitaetsmedizin Berlin /ID# 165186, Berlin
  - Helios Klinikum Wuppertal /ID# 165185, Wuppertal
- Japan (4):
  - Kurume University Hospital /ID# 165718, Kurume-shi, Fukuoka
  - Osaka General Medical Center /ID# 212745, Osaka, Osaka
  - Osaka University Hospital /ID# 165709, Suita-shi, Osaka
  - Juntendo University Hospital /ID# 212912, Bunkyo-ku, Tokyo
- San Jorge Children Hospital /ID# 160850, San Juan, Puerto Rico
- Russia (3):
  - Federal State Budgetary Institution - Institute of Nutrition /ID# 163345, Moscow, Moscow
  - National Medical Scientific Centre of children health /ID# 163344, Moscow, Moscow
  - Scientific and Research Institute of pediatric infections /ID# 163343, Saint Petersburg
- Spain (4):
  - Hospital Sant Joan de Deu /ID# 163282, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 163323, Barcelona
  - Hospital Universitario La Paz /ID# 163283, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 163325, Valencia
- United Kingdom (3):
  - Birmingham Childrens Hospital /ID# 162718, Birmingham
  - Queen Elizabeth University Hos /ID# 162719, Glasgow
  - King's College Hospital NHS /ID# 162717, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Jonas MM, Rhee S, Kelly DA, Del Valle-Segarra A, Feiterna-Sperling C, Gilmour S, Gonzalez-Peralta RP, Hierro L, Leung DH, Ling SC, Lobzin Y, Lobritto S, Mizuochi T, Narkewicz MR, Sabharwal V, Wen J, Kei Lon H, Marcinak J, Topp A, Tripathi R, Sokal E. Pharmacokinetics, Safety, and Efficacy of Glecaprevir/Pibrentasvir in Children With Chronic HCV: Part 2 of the DORA Study. Hepatology. 2021 Jul;74(1):19-27. doi: 10.1002/hep.31841. PMID 33811356
- [Derived] Jonas MM, Squires RH, Rhee SM, Lin CW, Bessho K, Feiterna-Sperling C, Hierro L, Kelly D, Ling SC, Strokova T, Del Valle-Segarra A, Lovell S, Liu W, Ng TI, Porcalla A, Gonzalez YS, Burroughs M, Sokal E. Pharmacokinetics, Safety, and Efficacy of Glecaprevir/Pibrentasvir in Adolescents With Chronic Hepatitis C Virus: Part 1 of the DORA Study. Hepatology. 2020 Feb;71(2):456-462. doi: 10.1002/hep.30840. Epub 2019 Aug 13. PMID 31254392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 38 sites in North America, Europe, and Japan. Cohort 1 enrolled adolescent participants aged 12 to < 18 years old. Subsequently, children aged 9 to < 12 (Cohort 2), 6 to < 9 (Cohort 3), and 3 to < 6 (Cohort 4) years old were enrolled in parallel.
Pre-assignment Details: In each cohort participants were first enrolled into an intense pharmacokinetic (IPK) portion to characterize the PK and safety, followed by a non-IPK safety/efficacy part. PK samples from the first 6 participants in the IPK part were analyzed to determine the final dose used for the remaining IPK participants and in the non-IPK group.
  A total of 129 participants were enrolled and 127 participants received at least 1 dose of study drug and were included in the intention-to-treat population.
Groups:
- Cohort 1: 12 to < 18 Years: Adolescents aged 12 to < 18 years old received the adult formulation of glecaprevir (GLE)/pibrentasvir (PIB) 100 mg/40 mg co-formulated film-coated tablets for a once daily (QD) total dose of 300 mg/120 mg by mouth for 8, 12, or 16 weeks depending on hepatitis C virus (HCV) genotype, cirrhosis status, and prior treatment experience.
- Cohort 2: 9 to < 12 Years: Children aged 9 to < 12 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 30 to < 45 kg was GLE 250 mg + PIB 100 mg.
- Cohort 3: 6 to < 9 Years: Children aged 6 to < 9 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 20 to < 30 kg was GLE 200 mg + PIB 80 mg; one participant received GLE 250 mg + PIB 100 mg based on weight at screening.
- Cohort 4: 3 to < 6 Years: Children aged 3 to < 6 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 12 to < 20 kg was GLE 150 mg + PIB 60 mg; one participant received GLE 200 mg + PIB 80 mg based on weight at screening.
Period: Overall Study
Arm/Group | Cohort 1: 12 to < 18 Years | Cohort 2: 9 to < 12 Years | Cohort 3: 6 to < 9 Years | Cohort 4: 3 to < 6 Years
Started | 47 | 29 | 27 | 24
Intense Pharmacokinetic Portion (Includes participants who provided IPK samples by age group) | 14 | 19 (Six participants received the initial proposed dose and 13 received the final proposed dose regimen.) | 18 (Six participants received the initial proposed dose and 12 received the final proposed dose regimen.) | 18 (Five participants received the initial proposed dose and 13 received the final proposed dose regimen.)
Completed | 42 | 24 | 22 | 18
Not Completed | 5 | 5 | 5 | 6
Not completed — Partially Dosed; Refused to Swallow Entire Dose | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 5 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population: all participants who received at least 1 dose of study drug
Groups:
- Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years: Adolescents aged 12 to < 18 years old received the adult formulation of glecaprevir (GLE)/pibrentasvir (PIB) 100 mg/40 mg co-formulated film-coated tablets for a once daily (QD) total dose of 300 mg/120 mg by mouth for 8, 12, or 16 weeks depending on hepatitis C virus (HCV) genotype, cirrhosis status, and prior treatment experience.
- Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years: Children aged 9 to < 12 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 30 to < 45 kg was GLE 250 mg + PIB 100 mg.
- Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years: Children aged 6 to < 9 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 20 to < 30 kg was GLE 200 mg + PIB 80 mg; one participant received GLE 250 mg + PIB 100 mg based on weight at screening.
- Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years: Children aged 3 to < 6 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 12 to < 20 kg was GLE 150 mg + PIB 60 mg; one participant received GLE 200 mg + PIB 80 mg based on weight at screening.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Total
Number analyzed (Participants) | 47 | 29 | 27 | 24 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.26 (1.51) | 10.00 (0.85) | 7.11 (0.89) | 3.79 (0.78) | 9.79 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 17 | 12 | 70
  Male | 21 | 14 | 10 | 12 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 4 | 4 | 18
  Not Hispanic or Latino | 42 | 24 | 23 | 20 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 21 | 18 | 16 | 90
  Black or African American | 4 | 1 | 1 | 1 | 7
  Asian | 6 | 5 | 5 | 4 | 20
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Multiple | 2 | 1 | 3 | 1 | 7
Baseline Fibrosis Stage [Count of Participants; unit: Participants] — Fibrosis stage was determined by biopsy score, FibroScan score (if biopsy not available), or FibroTest score (if biopsy and FibroScan not available) and is equivalent to the liver biopsy Metavir score:
  F0: no fibrosis; F1: portal fibrosis without septa; F2: portal fibrosis with few septa; F3: numerous septa without cirrhosis; F4: cirrhosis.
  Participants
    F0-F1 | 45 | 28 | 26 | 24 | 123
    F2 | 1 | 1 | 1 | 0 | 3
    F3 | 1 | 0 | 0 | 0 | 1
    F4 | 0 | 0 | 0 | 0 | 0
Hepatitis C Virus Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 37 | 19 | 22 | 17 | 95
  Genotype 2 | 3 | 2 | 0 | 0 | 5
  Genotype 3 | 4 | 8 | 3 | 7 | 22
  Genotype 4 | 3 | 0 | 2 | 0 | 5
  Genotype 5 | 0 | 0 | 0 | 0 | 0
  Genotype 6 | 0 | 0 | 0 | 0 | 0
Prior HCV Treatment History [Count of Participants; unit: Participants]
  Naive | 36 | 27 | 27 | 24 | 114
  Experienced | 11 | 2 | 0 | 0 | 13
Co-infection with Human Immunodeficiency Virus (HIV) [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 1 | 0 | 3
  No | 45 | 29 | 26 | 24 | 124
HCV Ribonucleic Acid (RNA) Level [Median (Full Range); unit: Log₁₀ IU/mL] — HCV RNA quantified by Roche COBAS Ampliprep/COBAS TaqMan HCV Quantitative Test, version 2.0.
  Log₁₀ IU/mL | 6.20 [4.63 to 7.18] | 6.20 [4.79 to 7.19] | 5.89 [4.53 to 7.15] | 5.83 [3.43 to 6.90] | 6.07 [3.43 to 7.19]

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC0-24) of Glecaprevir
Description: The area under the plasma concentration-time curve (AUC) is a method of measurement of the total exposure of a drug in blood plasma. The steady-state exposure of GLE was measured up to 24 hours after dosing at Week 2 and estimated using non-compartmental analysis.
Time Frame: Week 2 from predose to 24 hours post-dose
Population: Participants with intense pharmacokinetic samples who received the final dose regimen of GLE + PIB. One participant in Cohort 4 who received GLE 200 mg + PIB 80 mg based on weight (> 20 kg) is summarized in Cohort 3 for PK analyses based on the actual dose received.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Groups:
- Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years: Adolescents aged 12 to < 18 years old received the adult formulation of GLE/PIB 100 mg/40 mg co-formulated film-coated tablets for a once daily total dose of 300 mg/120 mg by mouth for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience.
- Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years: Children aged 6 to < 9 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 20 to < 30 kg was GLE 200 mg + PIB 80 mg.
- Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years: Children aged 3 to < 6 years old received a pediatric formulation of GLE + PIB as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience. The final dose for children weighing 12 to < 20 kg was GLE 150 mg + PIB 60 mg.
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years
Number analyzed (Participants) | 14 | 13 | 13 | 12
ng*h/mL | 4790 [3520 to 6500] | 7870 [4140 to 14900] | 6860 [4080 to 11500] | 7520 [3870 to 14600]

2. Primary Outcome: Steady-state AUC0-24 of Pibrentasvir
Description: The area under the plasma concentration-time curve (AUC) is a method of measurement of the total exposure of a drug in blood plasma. The steady-state exposure of PIB was measured up to 24 hours after dosing at Week 2 and estimated using non-compartmental analysis.
Time Frame: Week 2 from predose to 24 hours post-dose
Population: Participants with intense pharmacokinetic samples who received the final dose regimen of GLE + PIB. One participant in Cohort 4 who received GLE 200 mg + PIB 80 mg based on weight (> 20 kg) was summarized in Cohort 3 for PK analyses based on the actual dose received.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years
Number analyzed (Participants) | 14 | 13 | 13 | 12
ng*h/mL | 1380 [1150 to 1660] | 2200 [1460 to 3310] | 1640 [1230 to 2190] | 1790 [1350 to 2370]

3. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post Treatment (SVR12)
Description: SVR12 is defined as hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ; 15 IU/mL) 12 weeks after the last actual dose of study drug. Plasma HCV RNA levels were collected using the COBAS AmpliPrep/COBAS TaqMan HCV Quantitative Test v2.0.
  SVR12 was considered a primary efficacy endpoint by the United States (US) regulatory agency and was considered secondary outside of the US.
Time Frame: 12 weeks after last dose of study drug (Week 20, 24, or 28 depending on treatment duration)
Population: Intention-to-treat population: all participants who received at least 1 dose of study drug; Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backwards imputation were counted as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years: Children aged 3 to < 12 years old received a pediatric formulation of GLE + PIB at a final dose of GLE 250 mg + PIB 100 mg (children 9 to < 12 years of age), GLE 200 mg + PIB 80 mg (children 6 to < 9 years of age), or GLE 150 mg + PIB 60 mg (children 3 to < 6 years of age) as small film-coated granules taken with a small amount of food once daily for 8, 12, or 16 weeks depending on HCV genotype, cirrhosis status, and prior treatment experience.
- Total: Participants in Cohorts 1 to 4.
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years | Total
Number analyzed (Participants) | 47 | 29 | 27 | 24 | 80 | 127
percentage of participants | 100 [92.4 to 100.0] | 93.1 [78.0 to 98.1] | 100 [87.5 to 100.0] | 95.8 [79.8 to 99.3] | 96.3 [89.5 to 98.7] | 97.6 [93.3 to 99.2]

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Glecaprevir
Description: Cmax is the peak concentration that a drug or drug metabolite achieves in a specified compartment after the drug has been administered and before administration of a second dose.
Time Frame: Week 2 from predose to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years
Number analyzed (Participants) | 14 | 13 | 13 | 12
ng/mL | 1040 [733 to 1480] | 1370 [773 to 2440] | 1600 [926 to 2770] | 1530 [711 to 3290]

5. Secondary Outcome: Apparent Clearance (CL/F) of Glecaprevir From Plasma
Description: CL/F is a quantitative measure of the rate at which a drug substance is removed from the body. It was estimated by non-compartmental pharmacokinetic analysis.
Time Frame: Week 2 from predose to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/h
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years
Number analyzed (Participants) | 14 | 13 | 13 | 12
L/h | 62.6 [46.1 to 85.1] | 31.8 [16.7 to 60.3] | 29.1 [17.3 to 49.0] | 19.9 [10.2 to 38.7]

6. Secondary Outcome: Maximum Plasma Concentration of Pibrentasvir
Description: as for outcome 4
Time Frame: Week 2 from predose to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years
Number analyzed (Participants) | 14 | 13 | 13 | 12
ng/mL | 174 [148 to 205] | 225 [164 to 310] | 197 [154 to 251] | 233 [184 to 296]

7. Secondary Outcome: Apparent Clearance of Pibrentasvir From Plasma
Description: as for outcome 5
Time Frame: Week 2 from predose to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/h
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years
Number analyzed (Participants) | 14 | 13 | 13 | 12
L/h | 86.9 [72.4 to 104] | 45.4 [30.1 to 68.5] | 48.7 [36.6 to 64.8] | 33.6 [25.4 to 44.5]

8. Secondary Outcome: Percentage of Participants Who Experienced On-treatment Virologic Failure
Description: On-treatment virologic failure is defined as meeting one of the following:
  * A confirmed (defined as two consecutive HCV RNA measurements) increase of > 1 log₁₀ IU/mL above nadir during treatment;
  * Confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < 15 IU/mL during treatment;
  * HCV RNA ≥ 15 IU/mL at the end of treatment with at least 6 weeks of treatment.
Time Frame: Up to Week 8, 12, or 16 (depending on treatment duration)
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years | Total
Number analyzed (Participants) | 47 | 29 | 27 | 24 | 80 | 127
percentage of participants | 0 [0.0 to 7.6] | 0 [0.0 to 11.7] | 0 [0.0 to 12.5] | 0 [0.0 to 13.8] | 0 [0.0 to 4.6] | 0 [0.0 to 2.9]

9. Secondary Outcome: Percentage of Participants With Post-treatment Relapse up to 12 Weeks Post Treatment
Description: Post-treatment relapse is defined as confirmed HCV RNA ≥ 15 IU/mL between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment as planned with HCV RNA < 15 IU/mL at the end of treatment; excluding participants who had been shown to be re-infected.
Time Frame: Up to 12 weeks after the last dose of study drug (Week 20, 24, or 28 depending on treatment duration)
Population: Participants in the ITT population who completed treatment (based on study drug duration) with HCV RNA < 15 IU/mL at the final treatment visit and with at least one post-treatment HCV RNA value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years | Total
Number analyzed (Participants) | 47 | 28 | 27 | 23 | 78 | 125
percentage of participants | 0 [0.0 to 7.6] | 3.6 [0.6 to 17.7] | 0 [0.0 to 12.5] | 0 [0.0 to 14.3] | 1.3 [0.2 to 6.9] | 0.8 [0.1 to 4.4]

10. Secondary Outcome: Percentage of Participants With New Hepatitis C Virus Infection (Reinfection)
Description: Reinfection is defined as confirmed HCV RNA ≥ 15 IU/mL in the post-treatment period in a participant who had HCV RNA < 15 IU/mL at the Final Treatment Visit, along with post-treatment detection of a different HCV genotype, subtype, or clade compared with Baseline, as determined by phylogenetic analysis of the nonstructural viral protein 3 (NS3) or NS5A, and/or NS5B gene sequences.
Time Frame: From the end of treatment up to post-treatment Week 144
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years | Total
Number analyzed (Participants) | 47 | 29 | 27 | 24 | 80 | 127
percentage of participants | 0 [0.0 to 7.6] | 0 [0.0 to 11.7] | 0 [0.0 to 12.5] | 0 [0.0 to 13.8] | 0 [0.0 to 4.6] | 0 [0.0 to 2.9]

11. Secondary Outcome: Palatability Questionnaire Question 1: How Convenient or Inconvenient Was it to Prepare the Dose?
Description: For each participant who received the pediatric formulation (Cohorts 2 - 4), the parent(s)/guardian(s) completed a Palatability Questionnaire to provide feedback on the perception of the dosage form. The Palatability Questionnaire included 6 questions related to the administration and ingestion of the pediatric GLE + PIB formulation.
  Question 1 "How Convenient or Inconvenient Was it to Prepare the Dose?" was answered as "very convenient", "convenient", "borderline", "inconvenient", or "very inconvenient".
Time Frame: Final treatment visit (up to Week 8, 12, or 16, depending on treatment duration)
Population: Participants in the intention-to-treat population who completed the Palatability Questionnaire at the final treatment visit
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years
Number analyzed (Participants) | 28 | 27 | 23 | 78
Participants
  Very convenient | 7 | 9 | 9 | 25
  Convenient | 13 | 10 | 8 | 31
  Borderline | 2 | 7 | 4 | 13
  Inconvenient | 6 | 1 | 1 | 8
  Very inconvenient | 0 | 0 | 1 | 1

12. Secondary Outcome: Palatability Questionnaire Question 2: How Long Did it Typically Take for the Child to Take the Dose?
Description: For each participant who received the pediatric formulation (Cohorts 2 - 4), the parent(s)/guardian(s) completed a Palatability Questionnaire to provide feedback on the perception of the dosage form. The Palatability Questionnaire included 6 questions related to the administration and ingestion of the pediatric GLE + PIB formulation.
  Question 2 "How Long Did it Typically Take for the Child to Take the Dose?" was answered as "5 minutes or less", "5 to 15 minutes", "15 to 30 minutes", or "more than 30 minutes".
Time Frame: Final treatment visit (up to Week 8, 12, or 16, depending on duration of treatment)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years
Number analyzed (Participants) | 28 | 27 | 23 | 78
Participants
  5 minutes or less | 22 | 23 | 21 | 66
  5 to 15 minutes | 5 | 4 | 2 | 11
  15 to 30 minutes | 1 | 0 | 0 | 1
  More than 30 minutes | 0 | 0 | 0 | 0

13. Secondary Outcome: Palatability Questionnaire Question 3: Were You Able to Successfully Administer the Whole Dose to the Child With 1 to 2 Teaspoons (5 to 10 mL) of Soft Food?
Description: For each participant who received the pediatric formulation (Cohorts 2 - 4), the parent(s)/guardian(s) completed a Palatability Questionnaire to provide feedback on the perception of the dosage form. The Palatability Questionnaire included 6 questions related to the administration and ingestion of the pediatric GLE + PIB formulation.
  Question 3 "Were You Able to Successfully Administer the Whole Dose to the Child With 1 to 2 Teaspoons (5 to 10 mL) of Soft Food?" was answered as "Yes" or "No".
Time Frame: Final treatment visit (up to Week 8, 12, or 16, depending on treatment duration)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years
Number analyzed (Participants) | 28 | 27 | 23 | 78
Participants
  Yes | 20 | 19 | 19 | 58
  No | 8 | 8 | 3 | 19
  Missing | 0 | 0 | 1 | 1

14. Secondary Outcome: Palatability Questionnaire Question 4: Did You Experience Any Resistance When Feeding the Child the Medicine?
Description: For each participant who received the pediatric formulation (Cohorts 2 - 4), the parent(s)/guardian(s) completed a Palatability Questionnaire to provide feedback on the perception of the dosage form. The Palatability Questionnaire included 6 questions related to the administration and ingestion of the pediatric GLE + PIB formulation. Question 4 "Did You Experience Any Resistance When Feeding the Child the Medicine?" was answered as "Yes" or "No".
Time Frame: Final treatment visit (up to Week 8, 12, or 16 depending on treatment duration)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years
Number analyzed (Participants) | 28 | 27 | 23 | 78
Participants
  Yes | 6 | 4 | 7 | 17
  No | 22 | 23 | 15 | 60
  Missing | 0 | 0 | 1 | 1

15. Secondary Outcome: Palatability Questionnaire Question 4a: Type of Feeding Resistance
Description: For each participant who received the pediatric formulation (Cohorts 2 - 4), the parent(s)/guardian(s) completed a Palatability Questionnaire to provide feedback on the perception of the dosage form. The Palatability Questionnaire included 6 questions related to the administration and ingestion of the pediatric GLE + PIB formulation. Question 4a "Type of feeding resistance?" tracks feeding resistance experienced at any time during treatment, and was answered as "Did not like taste of medicine", "Did not like texture of medicine", "Did not like the soft food used", "Did not like to swallow the amount of medicine", or "Unrelated to the medicine".
Time Frame: Up to final treatment visit (up to Week 8, 12, or 16 depending on treatment duration)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years
Number analyzed (Participants) | 28 | 27 | 23 | 78
Participants
  Did not like taste of medicine | 3 | 5 | 6 | 14
  Did not like texture of medicine | 2 | 2 | 5 | 9
  Did not like the soft food used | 3 | 2 | 0 | 5
  Did not like to swallow the amount of medicine | 3 | 2 | 3 | 8
  Unrelated to the medicine | 0 | 0 | 1 | 1
  Missing | 0 | 0 | 1 | 1

16. Secondary Outcome: Palatability Questionnaire Question 5: How Easy or Difficult Was it for the Child to Swallow the Medicine?
Description: For each participant who received the pediatric formulation (Cohorts 2 - 4), the parent(s)/guardian(s) completed a Palatability Questionnaire to provide feedback on the perception of the dosage form. The Palatability Questionnaire included 6 questions related to the administration and ingestion of the pediatric GLE/PIB formulation. Question 5 "How Easy or Difficult Was it for the Child to Swallow the Medicine?" was answered as "very easy", "easy", "borderline", "difficult", or "very difficult."
Time Frame: Final treatment visit (up to Week 8, 12, or 16, depending on treatment duration)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years
Number analyzed (Participants) | 28 | 27 | 23 | 78
Participants
  Very easy | 10 | 8 | 11 | 29
  Easy | 13 | 16 | 10 | 39
  Borderline | 4 | 3 | 1 | 8
  Difficult | 1 | 0 | 0 | 1
  Very difficult | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study drug up to 30 days after last dose (up to 20 weeks depending on the duration of treatment). Deaths are reported through Post Treatment Week 144.
Arm/Group | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years | Total
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/29 | 0/27 | 0/24 | 0/80 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/29 | 0/27 | 0/24 | 0/80 | 0/127
Other Adverse Events (participants affected / at risk) | 31/47 | 15/29 | 16/27 | 17/24 | 48/80 | 79/127
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Adult Formulation GLE/PIB; 12 to < 18 Years (N=47) | Cohort 2: Pediatric Formulation GLE + PIB; 9 to < 12 Years (N=29) | Cohort 3: Pediatric Formulation GLE + PIB; 6 to < 9 Years (N=27) | Cohort 4: Pediatric Formulation GLE + PIB; 3 to < 6 Years (N=24) | Cohorts 2-4: Pediatric Formulation GLE + PIB; 3 to < 12 Years (N=80) | Total (N=127)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
MOTION SICKNESS (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 5 (6) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 2 (2) | 8 (8) | 11 (11)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 9 (9)
VOMITING (Gastrointestinal disorders) | 5 (5) | 1 (1) | 6 (6) | 4 (4) | 11 (11) | 16 (16)
FATIGUE (General disorders) | 5 (5) | 1 (1) | 3 (3) | 3 (3) | 7 (7) | 12 (12)
PYREXIA (General disorders) | 5 (6) | 1 (1) | 2 (3) | 2 (2) | 5 (6) | 10 (12)
LICE INFESTATION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 11 (12) | 4 (5) | 1 (1) | 1 (1) | 6 (7) | 17 (19)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (11) | 1 (1) | 3 (6) | 2 (2) | 6 (9) | 15 (20)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
HEADACHE (Nervous system disorders) | 8 (12) | 3 (3) | 6 (6) | 3 (3) | 12 (12) | 20 (24)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (6) | 7 (8) | 9 (10)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 3 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03067129/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT03067129/SAP_001.pdf